CLINICAL TRIAL: NCT03116412
Title: A Prospective Randomized Multicenter Trial to Assess the Role of Imaging During Follow Up After Radical Surgery of Stage IIb-c and III Cutaneous Malignant Melanoma
Brief Title: A Randomized Trial to Assess the Role of Imaging During Follow Up After Radical Surgery of High Risk Melanoma
Acronym: TRIM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Uppsala University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: TRIM
Record Dates: First submitted 2017-03-14; First posted 2017-04-17 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Malignant Melanoma
Keywords: Malignant melanoma; Follow up; Radiology; Survival
MeSH Terms: conditions — Melanoma | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Routine follow up (No Intervention): Follow up according to national guidelines.
- Radiological assessments (Experimental): Radiological assessments (CT or PET scans) at 5 occasions during 3 years.
  Interventions: Procedure: CT or PET scans

INTERVENTIONS:
Procedure: CT or PET scans — Scans and blood tests are scheduled at baseline, months 6, 12, 24 and 36.
  Arms: Radiological assessments

SUMMARY:
It is not known whether radiological assessments during follow up after surgery for high risk melanoma improve survival. Since radiological examinations are resource demanding, could inflict worry and cause irradiation exposure it is an important question to address. With the introduction of effective medical treatments for malignant melanoma patients, there is a tendency to introduce radiological assessments despite the lack of evidence.

DETAILED DESCRIPTION:
The patients are randomized 1:1 to routine follow up for 3 years with regular doctors´ appointments according to national guidelines and the same follow up but with the addition of whole body CT or Positron Emission Tomography (PET) scans and blood tests. An interim analysis will be conducted when 1000 patients have been included.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age.
* Radical surgery for Cutaneous Malignant Melanoma (CMM) stage IIb-c and III.
* Sufficient renal function for i.v. contrast scannings.

Exclusion Criteria:

* The patient is assessed as unfit to receive treatment in the case of recurrence.
* Life-expectancy less than 2 years due to concurrent disease (e.g., cardiac disease, terminal multiple sclerosis, liver cirrhosis).
* Inability to provide informed consent or refusal to do so.
* Inability to comply with the control or intense follow-up program.
* Participation in other clinical trials interfering with the control-program.
* Existing or previous malignancies within the past 5 years (except for in situ breast and cervical cancer, melanoma in situ and non-melanoma skin cancer).
* Pregnancy or currently planned pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1300 (Estimated)
Dates: Start 2017-06-08 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | At 5 years
  Measured from date of inclusion

SECONDARY OUTCOMES:
Quality of life/QLQ30 | During the 3 year intervention period
  Question of Life Questionnaire (QLQ) 30
Quality of life/HAD | During the 3 year intervention period
  Hospital, Anxiety and Depression (HAD) scale

OTHER OUTCOMES:
Disease free survival (DFS) | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Gustav Ullenhag, associate professor, Principal Investigator — Uppsala University Hospital
Locations (20):
- Sweden (20):
  - Södra Älvsborgs sjukhus, Borås
  - Mälarsjukhuset Eskilstuna, Eskilstuna
  - Falu lasarett, Falun
  - Gävle sjukhus, Gävle
  - Department of Surgery, Sahlgrenska University Hospital, Gothenburg
  - Helsingborgs lasarett, Helsingborg
  - Länssjukhuset Ryhov, Jönköping
  - Länssjukhuset i Kalmar, Kalmar
  - Centralsjukhuset i Karlstad, Karlstad
  - Linköping University Hospital, Linköping
  - Skåne University Hospital, Malmo
  - Örebro University Hospital, Örebro
  - Skaraborgs sjukhus Skövde, Skövde
  - Karolinska University Hospital, Stockholm
  - Länssjukhuset Sundsvall, Sundsvall
  - Uddevalla sjukhus, Uddevalla
  - Umeå University Hospital, Umeå
  - Akademiska sjukhuset, Uppsala
  - Västmanlands sjukhus Västerås, Västerås
  - Visby lasarett, Visby

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Ladjevardi CO, Naeser Y, Dyrke U, Papantoniou D, Bagge RO, Elander N, Ingvar C, Flygare P, Nilsson C, Jakobsson F, Lange-Norstrom K, Sundin A, Berglund A, Nyberg F, Ahringberg-Kald B, Helgadottir H, Ullenhag G. Physical examinations and whole-body imaging versus physical examinations alone during follow-up after radical surgery of stage IIB-C and III cutaneous malignant melanoma (TRIM): an interim analysis of a multicentre, randomised, phase 3 trial in Sweden. Lancet Oncol. 2025 Nov;26(11):1501-1510. doi: 10.1016/S1470-2045(25)00487-5. PMID 41167217
- [Derived] Naeser Y, Helgadottir H, Brandberg Y, Hansson J, Bagge RO, Elander NO, Ingvar C, Isaksson K, Flygare P, Nilsson C, Jakobsson F, Del Val Munoz O, Valachis A, Jansson M, Sparring C, Ohlsson L, Dyrke U, Papantoniou D, Sundin A, Ullenhag GJ. TRIM study protocol - a prospective randomized multicenter Trial to assess the Role of Imaging during follow-up after radical surgery of stage IIB-C and III cutaneous malignant Melanoma. BMC Cancer. 2020 Dec 7;20(1):1197. doi: 10.1186/s12885-020-07632-4. PMID 33287744